CLINICAL TRIAL: NCT00026637
Title: Depression and Health Outcomes in Refractory Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAB1084; 5R01NS040808-04 (NIH)
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Depression; Epilepsy
Keywords: depression; epilepsy; seizures
MeSH Terms: conditions — Depression; Epilepsy; Seizures | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sertraline (Active Comparator)
  Interventions: Drug: sertraline
- CBT (Active Comparator)
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Drug: sertraline — Sertraline: 25-200mg PO (orally); Subjects begin at 25mg for week 1 and increase to 50mg at the beginning of week 2. Sertraline is increased in 50mg increments when subjects score in the depressed range on the CES-D, a questionnaire that is administered every 2 weeks over the 16 week intervention period. Subjects may reduce dosage if toxicity occurs.
  Arms: Sertraline
Behavioral: cognitive behavior therapy — CBT (Cognitive Behavior Therapy) - CBT is a psychotherapy based on modifying cognitions, assumptions, beliefs and behaviors, with the aim of influencing disturbed emotions. Subjects will meet with a trained CBT therapist for 1 hour each week over the 16 week intervention period and will be given assignments to work on each week.
  Other Names: CBT
  Arms: CBT

SUMMARY:
To define the benefits of antidepressant treatment or cognitive behavior therapy on mood, function, and quality of life in persons with depression and refractory epilepsy.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted to compare the drug sertraline to cognitive behavioral therapy on symptoms of depression, antiepileptic medication compliance, seizure frequency, and quality of life outcomes in persons with depression and a seizure disorder or epilepsy. Approximately 140 persons will be enrolled in this study over a period of five years. Individual participation will last approximately 16 weeks. Study participants will be chosen randomly to receive either the study medication (sertraline) or cognitive behavior therapy for 16 weeks. Sertraline is approved by the Food and Drug Administration (FDA). Subjects who receive cognitive behavior therapy will be provided with a one-hour individual session with a licensed clinical psychologist each week for 15 weeks. All study participants will attend scheduled clinic visits every 4 weeks for 16 weeks.

ELIGIBILITY:
INCLUSION:

* Must have a seizure disorder.
* Must meet the DSM-IV criteria for major depression.
* Must be willing to provide written informed consent.
* Must be age 21 to 75 years old.
* Must be compliant, cooperative, reliable, and able to follow instructions, and to visit the clinic on schedule.

EXCLUSION:

* Have active suicidal or homicidal ideation.
* Have current alcohol or other substance abuse disorders or a history of bipolar depression or any psychotic disorder.
* Are pregnant or lactating.
* Are known to be hypersensitive to sertraline.
* Have a progressive central nervous system disorder (such as a tumor or multiple sclerosis), or severe hepatic or renal disease (serum creatinine >3 mg/dl).
* Currently taking an antidepressant medication or seeing a therapist regularly.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2001-08; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
MINI | completed at screen and 16 weeks

SECONDARY OUTCOMES:
Depression as measured by the CES-D | completed every 2 weeks during the 16 week intervention period and at 6 month and 1 year follow ups
Health Related Quality of life as measured by the QOILIE-89 | completed every 4 weeks during the 16 week intervention period and at 6 month and 1 year follow ups
antiepileptic medication compliance | assessed at 16 weeks
antiepileptic medication toxicity as measured by the AEP | assessed every 2 weeks during the 16 week intervention period
seizure frequency and seizure severity | assessed every 2 weeks during the 16 week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gilliam, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maguire MJ, Marson AG, Nevitt SJ. Antidepressants for people with epilepsy and depression. Cochrane Database Syst Rev. 2021 Apr 16;4(4):CD010682. doi: 10.1002/14651858.CD010682.pub3. PMID 33860531